CLINICAL TRIAL: NCT02364960
Title: Implementation of the Target Intraoperative Therapy Registry at Bethesda North TriHealth Hospital (TARGIT)
Brief Title: Targeted Intraoperative Therapy Registry at Bethesda North Hospital (TARGIT)
Acronym: TARGIT
Status: Terminated | Type: Observational
Why Stopped: Study site will join the TARGIT-US trial in lieu of this trial
Sponsor: TriHealth Inc. (Other)
Collaborators: TriHealth Hatton Research Institute (Other); Bethesda North Hospital Foundation (Unknown)
Responsible Party: Principal Investigator, Angela N Fellner PhD CCRP, Co-Director, Mary Jo Cropper Family Center for Breast Care, TriHealth Inc.
Other Study IDs: 14-047
Record Dates: First submitted 2015-01-26; First posted 2015-02-18 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Early Stage Breast Cancer; Neoplasm of the Breast; Breast Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create a registry to evaluate the use of intra-operative radiation therapy (IORT) and to study the efficacy and toxicity of breast radiotherapy given intra-operatively as a single fraction after breast conserving surgery,

DETAILED DESCRIPTION:
A registry trial has been designed and modeled after the original successful TARGIT protocol, to continue the use of IORT for a select population of women, and to follow outcomes with regards to local and regional control, toxicity and morbidity. Patients selected for breast conserving surgery, who are considered to have a low risk of local recurrence, are eligible for this registry trial once their informed consent is obtained. This single arm cohort study allows entry of patients who have been diagnosed with early stage breast cancer and whose clinical stage is suitable for treating conservatively (small tumor and no gross nodal involvement). Tumors should not be more than 3.5 cm in size.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 45 or greater
* Diagnosed with operable invasive breast cancer, T1 and T2 (< 3.5 cm), N0, M0, confirmed by cytological or histological examination
* Suited for breast conserving surgery
* Have had an ipsilateral (same side as current cancer) diagnostic mammogram within 12 months of enrollment

Exclusion Criteria:

* age 44 or less
* Axillary lymph node positive breast cancer
* Invasive lobular cancer
* Tumor size > 3.5 cm
* Extensive Intraductal Component (EIC= > 25% of the lumpectomy specimen involved with ductal carcinoma in situ, DCIS) as assessed on surgical pathologic lumpectomy specimen
* Multicentric cancer in the same breast not amenable to excision with a single lumpectomy
* Inability to assess pathologic margin status
* Synchronous bilateral breast cancer at the time of diagnosis.
* Ipsilateral breast had a previous cancer and/or prior in-field radiation.
* Patients known to have BRCA1/2 gene mutations
* Neoadjuvant treatment (hormones or chemotherapy)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, aged 45 and greater who have been diagnosed with early stage invasive breast cancer that is suitable for breast conserving surgery.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
In-breast local failure and patterns of in-breast failure | 6 months after IORT through year 10
  In-breast local failure is defined as recurrence of cancer in the ipsilateral (same side) breast. Following IORT, patients will be monitored every 6 months for 3 years, and then annually in years 4 and 5 to determine if cancer has returned. In years 6 through 10 medical records will be reviewed to obtain information on participants' breast cancer status.

CONTACTS AND LOCATIONS:
Overall Officials: Ching Ho, MD PhD, Principal Investigator — Mary Jo Cropper Family Center for Breast Care
Locations (1):
- Mary Jo Cropper Family Center for Breast Care, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No